CLINICAL TRIAL: NCT07216274
Title: Quantitative Transmission Imaging Evaluation (QTIE Study) Compared With MRI as Supplemental Screening in Patients With High Lifetime Risk of Breast Cancer
Brief Title: Quantitative Transmission Imaging Compared With MRI as Supplemental Screening for High Lifetime Risk of Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 24-008575; NCI-2025-07168 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-008575 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2025-10-08; First posted 2025-10-14 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Screening (QTI) (Experimental): Patients undergo QTI ultrasound imaging on study.
  Interventions: Device: QT Ultrasound Breast Scanner; Other: Questionnaire Administration

INTERVENTIONS:
Device: QT Ultrasound Breast Scanner — Undergo Quantitative Transmission Imaging (QTI) using the QT Ultrasound Breast Scanner
  Other Names: 3D ultrasound; QTI; QT Ultrasound; Quantitative Transmission Ultrasound (QTUS); Quantitative Transmission Imaging
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial compares the use of quantitative transmission imaging (QTI) to standard of care MRI as a supplemental screening tool for patients with a high lifetime risk of breast cancer. QTI is a single 3D ultrasound test intended to be used as an initial evaluation method for asymptomatic women identified with above-average risk for developing breast cancer. Using QTI may be an effective supplemental screening tool, compared to MRI for patients with a high lifetime risk of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women 18+ years of age
* High lifetime risk of breast cancer as determined by a risk assessment tool such a Tyrer-Cuzick model
* Clinical ordered screening MRI.

  * MRI and QTI performed within 30 days of each other
* Breasts that will fit in the quantitate transmission (QT) Ultrasound Breast Scanner (e.g. bra cup size less than DDD)

Exclusion Criteria:

* Pregnant patients
* Lactating patients
* Patients with open wounds or discharge
* Patients < 18 years of age
* Patients who are > 350 lbs
* Patients who are unable to lay prone for >15 minutes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2025-07-31 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Detectability of positive exam findings (feasibility) | Baseline
  Assessed by description of the number of positive findings. Breast Imaging Reporting and Data System (BIRADS) classification of the screening exam and potential diagnostic work up may allow for calculation of positive predictive value (PPV)1 and PPV3. If biopsies are obtained, then findings will be compared to histopathologic diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany M. Sae-Kho, MD, Principal Investigator — Mayo Clinic in Rochester; Christine U. Lee, MD, PhD, Principal Investigator — Mayo Clinic in Rochester; Chidi T. Nwachukwu, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials